CLINICAL TRIAL: NCT02566720
Title: Mechanism of Amantadine and Functional Improvement Following Acquired Brain Injury as Measured by MRI Tractography; A Pilot Study
Brief Title: Amantadine and Functional Improvement Following ABI Measured by MRI Tractography; A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0452
Record Dates: First submitted 2015-09-23; First posted 2015-10-02 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Acquired Brain Injury; Coma; Persistent Vegetative State; Minimally Conscious State; Traumatic Brain Injury
Keywords: amantadine; tractography; mri; coma; abi; tbi; traumatic brain injury; acquired brain injury
MeSH Terms: conditions — Brain Injuries; Coma; Persistent Vegetative State; Brain Injuries, Traumatic | interventions — Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment and MRI scanning (Other): After informed consent has been obtained, the subjects will be examined by a physician and assigned a Disability Ratings Scale (DRS) score. Subjects will undergo MRI tractography study, which does not require the administration of contrast. All participants will receive oral amantadine at escalating doses to ensure tolerance (50mg twice daily for 7 days, then 100mg twice daily for 1 week, then 150mg twice daily, then 200mg twice daily). The usual length of stay on the inpatient brain injury program is ninety days. The MRI tractography study and DRS score will be repeated near the time of discharge or ninety days from enrollment.
  Interventions: Drug: Amantadine; Procedure: MRI Tractography Study

INTERVENTIONS:
Drug: Amantadine — Participants will initially receive amantadine at the starting dose of 50mg twice daily either by mouth or feeding tube. The dosage will increase every week by 50mg twice daily (100mg total dose increase) up to the target dose of 200mg twice daily. These are the usual doses and rate of increase that are offered to patients with brain injury.
  Other Names: amantadine hydrochloride
Procedure: MRI Tractography Study — Participants will initially receive a baseline MRI Tractography scan. The size of RAS fiber tracts will be measured prior to initiating treatment and near the time of discharge from the rehabilitation hospital or at approximately ninety-days.

SUMMARY:
This is a pilot study. The objective is to further understand the mechanism by which amantadine improves function in patients with persistent vegetative state and minimally conscious state. Specifically, the investigators will measure the size of the nerve fibers that mediate arousal (reticular activating system, or RAS) pre and post treatment on MRI tractography. MRI findings will be correlated with the Disability Rating Scale (DRS) score. The information gathered from this study will be used to formulate a larger clinical trial.

DETAILED DESCRIPTION:
Primary Aim:

To determine the size of the RAS tracts as measured by MRI tractography. Specifically, the investigators will be measuring the fiber tracts that project through the posterior thalamus. The RAS is involved in mediating arousal and consciousness. The size of fiber tracts will be measured prior to initiating treatment and near the time of discharge from the rehabilitation hospital or at approximately ninety-days. It is hypothesized that treatment will result in an increase in the size of these fiber tracts.

As a pilot study, the investigators will be determining the feasibility of recruiting and retaining patients in this type of study. This will allow the clarification and understanding of the technical standards for MRI tractography related to the assessment of the reticular activating system.

Secondary Aim:

To determine and monitor changes in function following acquired brain injury as measured by the Disability Rating Scale (DRS) score. The DRS score will be obtained prior to initiating treatment and at termination of the study. It is hypothesized that treatment with amantadine in addition to standard medical treatment, will be associated with an improvement in function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years - 65 years
* Nonpenetrating acquired brain injury (ABI)
* Persistent vegetative or minimally conscious state (as indicated by DRS score greater than 11)
* Consent from substitute decision maker

Exclusion Criteria:

* Contraindication to MRI (such as metal in the body, pacemaker, implanted nerve stimulator)
* Anticipated neurosurgical intervention
* Medical instability including uncontrolled hypertension, fever, or infection
* Seizure disorder prior to acquired brain injury or uncontrolled seizures subsequent to acquired brain injury
* Parkinson's disease
* History of heart failure or pre-existing peripheral oedema
* History of eczematoid dermatitis
* History of angle-closure glaucoma
* History of neuroleptic malignant syndrome
* Current treatment with Amantadine
* Impairment related to other neurologic disease other than ABI
* Allergy to Amantadine
* Pregnancy or lactation
* Impairment of renal function (creatinine clearance less than 60ml/min)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Radiographic Changes | At baseline and ninety days or at time of discharge from hospital if occurs earlier.
  MRI Tractography will be performed to measure the size the of reticular activating system fiber tracts. Specifically, the tracts that project through the posterior thalamus.

SECONDARY OUTCOMES:
Functional Improvement | At ninety days or at time of discharge from hospital if occurs earlier.
  Disability Rating Scale Score (at enrolment and at completion of the study).

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj E Bansal, MD, Principal Investigator — Hamilton Health Sciences Corporation; Seyed Hosseini, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada